CLINICAL TRIAL: NCT04838262
Title: Daily Stress Processes and Sympathetic Reactivity in Depression
Brief Title: Stress and the Sympathetic Nervous System in Adults With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: Penn State University (Other)
Responsible Party: Principal Investigator, Jody Greaney, Principal Investigator, University of Delaware
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MH123928
Record Dates: First submitted 2021-03-31; First posted 2021-04-09 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessment of Daily Stress Processes (Experimental): Subjects will report cumulative exposure, perceived severity, and emotional responsiveness to commonly occurring everyday psychosocial stressors utilizing an ecological momentary assessment approach for 8 consecutive days.
  Interventions: Other: Acute Stressors

INTERVENTIONS:
Other: Acute Stressors — Sympathetic nervous system activity and blood pressure will be measured before, during, and after several acute laboratory-based cognitive (Stroop Color Word Test), emotional (International Affective Picture System), and physiological (Cold Pressor Test) stressors.

SUMMARY:
To test our hypotheses, we will enroll healthy adults having no history of mood disorders and adults with major depressive disorder (MDD) having a broad range of depressive symptom severity. After screening, subjects will meet with the research coordinator or an investigator for a discussion, with opportunity for questions, before applicable consent forms are obtained. Daily stress processes will be assessed using an ecological momentary assessment approach for 8 consecutive days. On the last day of the daily stress assessment, we will directly measure muscle sympathetic nerve activity, blood pressure, and heart rate during acute laboratory-based cognitive, emotional, and physiological interventions to induce a stress response. A venous blood sample will be taken for measurements of metabolic and renal health and systemic inflammation.

Aim 1: To examine the effect of daily psychosocial stressor exposure on acute sympathetic stress reactivity in MDD. Two stressor exposure indicators will be calculated: stressor frequency (i.e., percentage of interview days during which at least one stressor occurred) and total stress (i.e., total number of stressors reported across all interview days) and will be related to the magnitude of responsiveness to the acute stress interventions. We hypothesize that the slope of this relation will be steeper in adults with MDD compared to healthy non-depressed adults.

Aim 2: To determine the relation between negative affective reactivity to daily psychosocial stressor exposure and acute sympathetic stress reactivity in MDD. Negative affective reactivity will be calculated as the change in affect on days when stressors occurred compared to one's typical affect on non-stressor days and will be related to the magnitude of responsiveness to the acute stress interventions. We hypothesize that the slope of this relation will be steeper in adults with MDD compared to healthy non-depressed adults.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be 18-30 yrs.
* Healthy non-depressed men and women will have no history or evidence of psychiatric illness and will not have a family history of MDD or major psychiatric illness.
* Men and women with MDD will have symptomatic depression that meets diagnostic criteria and will be non-medicated.
* The capacity and willingness to provide written informed consent, to attend all study related visits, and to comply with the study protocol.

Exclusion Criteria:

Subjects will be excluded at the discretion of the PI/collaborating clinician or for any of the following reasons:

* psychiatric illness aside from MDD (including current or past psychotic disorders, bipolar disorder, schizophrenia or schizoaffective disorder, panic disorder, post-traumatic stress disorder, obsessive compulsive disorder)
* subthreshold depression
* current use of psychotropic medications (including major classes of antidepressants, anxiolytics, antipsychotics, mood stabilizers)
* active suicidal or homicidal ideation
* active substance dependence or eating disorders
* current use of any medications that could alter sympathetic reactivity
* diagnosed or suspected cardiovascular, renal, or metabolic disease (hypertension, heart disease, diabetes, hyperlipidemia)
* autonomic disorders
* tobacco use (including electronic cigarettes)
* obesity (body mass index > 30 kg/m2)
* breastfeeding or pregnancy
* <18 or >30 yrs

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Arlington, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Per the data sharing policy of the National Institute of Mental Health (NIMH), we will deposit all phenotypic, psychosocial stress, and sympathetic reactivity data from this study to the NIMH Data Archive. We will use standard data dictionaries (NIH Toolbox Cognition Battery, NIH Toolbox Emotion Battery, Patient Health Questionnaire (PHQ)-9) and will collect the data necessary to generate global unique identifiers for each study subject.

REFERENCES:
- [Derived] Darling AM, Young BE, Skow RJ, Dominguez CM, Saunders EFH, Fadel PJ, Greaney JL. Sympathetic and blood pressure reactivity in young adults with major depressive disorder. J Affect Disord. 2024 Sep 15;361:322-332. doi: 10.1016/j.jad.2024.06.053. Epub 2024 Jun 17. PMID 38897296

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This protocol was registered and approved as a Single Arm/Group Assignment Intervention Model, consistent with the description in the associated funded grant. All participants received the same intervention. Data are reported separately for each group (HA, MDD); however, the influence of depression on the outcome variables was determined statistically by the presence of a significant interaction term in the model when combining Arm/Group.
Groups:
- Non-depressed Healthy Adults (HA): HA had no history or evidence of psychiatric illness and had no family history of MDD or major psychiatric illness.
  HA reported cumulative exposure, perceived severity, and emotional responsiveness to commonly occurring everyday psychosocial stressors utilizing an ecological momentary assessment approach for 8 consecutive days. Sympathetic nervous system activity and blood pressure were measured before, during, and after several acute laboratory-based cognitive (Stroop Color Word Test), emotional (International Affective Picture System), and physiological (Cold Pressor Test) stressors.
- Adults With Major Depressive Disorder (MDD): Adults with MDD had symptomatic depression that met diagnostic criteria and were not medicated.
  Adults with MDD reported cumulative exposure, perceived severity, and emotional responsiveness to commonly occurring everyday psychosocial stressors utilizing an ecological momentary assessment approach for 8 consecutive days. Sympathetic nervous system activity and blood pressure were measured before, during, and after several acute laboratory-based cognitive (Stroop Color Word Test), emotional (International Affective Picture System), and physiological (Cold Pressor Test) stressors.
Period: Overall Study
Arm/Group | Non-depressed Healthy Adults (HA) | Adults With Major Depressive Disorder (MDD)
Started | 51 | 43
Completed | 42 | 39
Not Completed | 9 | 4
Not completed — Withdrawal by Subject | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-depressed Healthy Adults (HA) | Adults With Major Depressive Disorder (MDD) | Total
Number analyzed (Participants) | 42 | 39 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 39 | 81
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22 (4) | 22 (5) | 22 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 31 | 58
  Male | 15 | 8 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 16 | 29
  Not Hispanic or Latino | 29 | 23 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 5 | 8
  Asian | 15 | 13 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 16 | 18 | 34
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 39 | 81
Patient Health Questionnaire (PHQ)-9 [Mean (Standard Deviation); unit: arbitrary units] — Patient Health Questionnaire-9 (PHQ-9) severity measure for depression. Total score reported on possible range of 0 to 27. The minimal score of 0 indicates the absence of depressive symptoms. The maximal score of 27 indicates the presence of the most severe depressive symptoms.
  arbitrary units | 3.1 (2.9) | 7.9 (5.4) | 5.4 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Days Participants Report Stressors
Description: the percentage of days that participants reported stressors over the course of 8 days before the intervention, measured each day via self-report using ecological momentary assessment
Time Frame: 8 days before intervention
Population: This protocol was registered and approved as a Single Arm/Group Assignment Intervention Model, consistent with the description in the associated funded grant. All participants received the same intervention. Data are reported separately for each group (HA, MDD); however, the influence of depression on the outcome variables was determined statistically by the presence of a significant interaction term in the model when combining Arm/Group.
Measure: Mean (Standard Deviation); unit: percent of days
Arm/Group | Non-depressed Healthy Adults (HA) | Adults With Major Depressive Disorder (MDD)
Number analyzed (Participants) | 42 | 39
percent of days | 36 (26) | 40 (24)

2. Primary Outcome: Negative Affective Reactivity to Daily Stressors
Description: Negative affect was measured each day via self-report using ecological momentary assessment using Positive and Negative Affect Schedule (possible range 1-5 arbitrary units, AU), and negative affective reactivity score was defined as the magnitude of the change in negative affect on days when stressors occurred compared to negative affect on non-stressor days over the 8-day timeframe. A singe negative affective reactivity score was calculated for each participant using two-level multi-level modeling (within person slopes). This outcome was operationalized as described in the funded grant and does not have a scale/construct name. There is no defined/set range: more negative slopes indicate a paradoxical increase in negative affect on stressor days, whereas more positive slopes indicate a greater decline in negative affect on stressor days.
Time Frame: 8 days before intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: AU stressor days/AU non-stressor days
Arm/Group | Non-depressed Healthy Adults (HA) | Adults With Major Depressive Disorder (MDD)
Number analyzed (Participants) | 42 | 39
AU stressor days/AU non-stressor days | 0.24 (0.08) | 0.31 (0.10)

3. Primary Outcome: Change in Muscle Sympathetic Nerve Activity in Response to Acute Stress (Compared to Resting Baseline Activity)
Description: muscle sympathetic nerve activity was measured using microneurography and the change was calculated as the difference between the mean value during baseline and during the mean value during each of three laboratory-based interventions (cold pressor test, Stroop color word test, International Affective Picture System); a larger value indicates a greater increase in sympathetic activity
Time Frame: 3 minutes after each laboratory-based intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bursts per minute
Arm/Group | Non-depressed Healthy Adults (HA) | Adults With Major Depressive Disorder (MDD)
Number analyzed (Participants) | 42 | 39
bursts per minute
  cold pressor test | 24.1 (12.0) | 21.4 (10.9)
  Stroop color word test | -2.3 (6.9) | -2.6 (6.5)
  International Affective Picture System | 0.8 (3.7) | 2.3 (4.8)
Statistical Analysis 1: Comparison: Non-depressed Healthy Adults (HA) vs Adults With Major Depressive Disorder (MDD); Test type: Other; p = 0.57, Regression, Linear
Statistical Analysis 2: Comparison: Non-depressed Healthy Adults (HA) vs Adults With Major Depressive Disorder (MDD); Test type: Other; p = 0.85, Regression, Linear

ADVERSE EVENTS:
Time Frame: 8 days
Arm/Group | Non-depressed Healthy Adults (HA) | Adults With Major Depressive Disorder (MDD)
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/43
Other Adverse Events (participants affected / at risk) | 0/51 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT04838262/Prot_001.pdf
  • Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT04838262/SAP_002.pdf
  • Informed Consent Form (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT04838262/ICF_000.pdf